CLINICAL TRIAL: NCT05162469
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of SHR-1909 Injection in Patients With Advanced Malignant Tumors
Brief Title: A Study of SHR-A1909 in Subjects With Advanced Malignant Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1909-I-101
Record Dates: First submitted 2021-12-05; First posted 2021-12-17 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Advanced Malignant Cancer

STUDY DESIGN:
Intervention Model Description: Dose escalation (non randomized， 6 arms); Dose-expansion and efficacy-expansion(non-randomized,1-3 arms)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1909 monotherapy (Experimental)
  Interventions: Drug: SHR-1909 injection

INTERVENTIONS:
Drug: SHR-1909 injection — SHR-1909 for intravenous injection;Strength:6ml:0.3g/vial. Dose escalation (non randomized, 6 dose-levels); Dose-expansion and efficacy-expansion(non-randomized,1-3 dose-level(s)).

SUMMARY:
This is an, open-label, multi-center, three-part phase I trial to evaluate the safety, pharmacokinetics and immunogenicity of SHR-1909 and preliminary anti-tumor efficacy of SHR-1909 in advanced malignant cancer.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Patients must have cytologically or histologically confirmed advanced malignant tumor, and must have failed standard treatment;
* Toxicities caused by prior anti-tumor treatments must have resolved to CTCAE Grade ≤ 1 prior to the first dose (except for alopecia or hypothyroidism treated with hormone replacement therapy or diabetes controlled with insulin);
* Adequate organ function.

Exclusion Criteria:

* With CNS infiltration, or ascites requiring paracentesis or symptomatic pleural effusion;
* Received prior CAR T-cell therapy;
* Received allogeneic hematopoietic stem cell transplantation within 3 months prior to the start of study treatment, or with acute/chronic graft versus host disease;
* With active infection or fever of unknown origin (> 38.5 °C).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
MTD of SHR-1909 | From Day 1 to 4 weeks
  Maximum tolerated dose (MTD) based on dose-limiting toxicities (DLTs)
RP2D of SHR-1909 | From Day 1 to 90 days after last dose
  Recommended Phase 2 Dose(RP2D) of SHR-1909 will be determined during the dose-escalation and dose-expansion parts of the study. RP2D will be determined using available safety, pharmacokinetics and pharmacodynamics data.

SECONDARY OUTCOMES:
Adverse Events | 90 days after the last dose
  Adverse Events documented by CTCAE 5.0
Objective Response Rate (ORR) | Up to approximately 2 years
  Baseline to documented disease progression or study discontinuation
Progression-Free Survival (PFS) | Up to approximately 2 years
  From Day 1 to Radiographic Progression or Death Due to Any Cause

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin Cancer Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided